CLINICAL TRIAL: NCT05194592
Title: Comparison of the Effects of Dapagliflozin and Gemigliptin on Ketone Metabolism and Cardiac Remodeling in Type 2 Diabetes
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wonju Severance Christian Hospital (Other)
Responsible Party: Principal Investigator, Dong-Hyuk Cho, Assistant Professor, Wonju Severance Christian Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR121038
Record Dates: First submitted 2022-01-04; First posted 2022-01-18 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Type2 Diabetes; Remodeling, Ventricular
MeSH Terms: conditions — Ventricular Remodeling | interventions — dapagliflozin; LC15-0444

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dapagliflozin group (Active Comparator): Dapagliflozin 10mg for 6 months.
  Interventions: Drug: Dapagliflozin
- Gemigliptin group (Placebo Comparator): Gemigliptin 50mg for 6 months.
  Interventions: Drug: Gemigliptin

INTERVENTIONS:
Drug: Dapagliflozin — The patients assigned to the Dapagliflozin group will take Farxiga Pill 10mg for 6 months.
  Arms: Dapagliflozin group
Drug: Gemigliptin — The patients assigned to the Gemigliptin group will take Zemiglo Pill 50mg for 6 months.
  Arms: Gemigliptin group

SUMMARY:
Sodium-glucose cotransporter 2 (SGLT2) inhibitors have demonstrated cardiovascular and renal protection in patients with type 2 diabetes (T2D); however, the underlying mechanism remains unclear. We hypothesized that SGLT2 inhibitor will improve the ketone metabolism compared to dipeptidyl Peptidase-4 (DPP4) inhibitor. And we will also evaluate the association between ketone metabolism and cardiac remodeling evaluated by echocardiography. We will randomly assign 122 people with T2DM to receive dapagliflozin 10mg or gemigliptin 50mg. The primary endpoint are changes in acetoacetate, total ketone, beta-hydroxybutyric acid, left ventricular (LV) mass index, and LV global longitudinal strain during 6 months follow-up. This study may provide robust evidence of the thrifty substrate hypothesis for cardiovascular protection of SGLT2 inhibitors.

ELIGIBILITY:
Inclusion Criteria:

* Subjects diagnosed with T2D on stable antidiabetic medication
* No recent use of SGLT2 inhibitor within 3 months

Exclusion Criteria:

* HbA1c > 10%
* Pregnancy or breast feeding
* estimated GFR <45 30 mL/min/1.73㎡
* insulin user

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Estimated)
Dates: Start 2022-01-07 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Change (%) in acetoacetate, total ketone, beta-hydroxybutyric acid | 6 months
  The change of acetoacetate, total ketone, beta-hydroxybutyric acid from baseline to 6 months follow-up
Change (%) in LV mass index | 6 months
  The change of LV mass index from baseline to 6 months follow-up

SECONDARY OUTCOMES:
Change (%) in LV ejection global longitudinal strain | 6 months
  The change of LV mass ejection global longitudinal strain from baseline to 6 months follow-up
Change (%) in mean 24hr ambulatory systolic and diastolic blood pressure | 6 months
  The change of mean 24hr ambulatory systolic and diastolic blood pressurefrom baseline to 6 months follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Yonsei University Wonju College of Medicine, Wŏnju, Gangwondo, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Correction. J Am Coll Cardiol. 2020 Sep 22;76(12):1505. doi: 10.1016/j.jacc.2020.08.010. No abstract available. PMID 32943171
- [Background] Tikkanen I, Narko K, Zeller C, Green A, Salsali A, Broedl UC, Woerle HJ; EMPA-REG BP Investigators. Empagliflozin reduces blood pressure in patients with type 2 diabetes and hypertension. Diabetes Care. 2015 Mar;38(3):420-8. doi: 10.2337/dc14-1096. Epub 2014 Sep 30. PMID 25271206
- [Background] Verma S, McMurray JJV. SGLT2 inhibitors and mechanisms of cardiovascular benefit: a state-of-the-art review. Diabetologia. 2018 Oct;61(10):2108-2117. doi: 10.1007/s00125-018-4670-7. Epub 2018 Aug 22. PMID 30132036
- [Background] Kim SR, Lee SG, Kim SH, Kim JH, Choi E, Cho W, Rim JH, Hwang I, Lee CJ, Lee M, Oh CM, Jeon JY, Gee HY, Kim JH, Lee BW, Kang ES, Cha BS, Lee MS, Yu JW, Cho JW, Kim JS, Lee YH. SGLT2 inhibition modulates NLRP3 inflammasome activity via ketones and insulin in diabetes with cardiovascular disease. Nat Commun. 2020 May 1;11(1):2127. doi: 10.1038/s41467-020-15983-6. PMID 32358544
- [Background] Gaborit B, Ancel P, Abdullah AE, Maurice F, Abdesselam I, Calen A, Soghomonian A, Houssays M, Varlet I, Eisinger M, Lasbleiz A, Peiretti F, Bornet CE, Lefur Y, Pini L, Rapacchi S, Bernard M, Resseguier N, Darmon P, Kober F, Dutour A. Effect of empagliflozin on ectopic fat stores and myocardial energetics in type 2 diabetes: the EMPACEF study. Cardiovasc Diabetol. 2021 Mar 1;20(1):57. doi: 10.1186/s12933-021-01237-2. PMID 33648515
- [Background] Brown AJM, Gandy S, McCrimmon R, Houston JG, Struthers AD, Lang CC. A randomized controlled trial of dapagliflozin on left ventricular hypertrophy in people with type two diabetes: the DAPA-LVH trial. Eur Heart J. 2020 Sep 21;41(36):3421-3432. doi: 10.1093/eurheartj/ehaa419. PMID 32578850